CLINICAL TRIAL: NCT04335383
Title: Isolation of Human Recombinant Therapeutic Monoclonal Anti-Pseudomonas Antibodies From B Lymphocytes of Patients Who Have Been Followed for Infection or Colonization With Pseudomonas Aeruginosa: a Prospective Monocentric Trial
Brief Title: Isolation of Human Recombinant Therapeutic Monoclonal Anti-Pseudomonas Antibodies
Acronym: ABAC-IBS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.048; 2020-A00311-38 (Other: ID RCB)
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Pseudomonas Aeruginosa; Multi-antibiotic Resistance
Keywords: Pseudomonas aeruginosa; monoclonal antibody
MeSH Terms: conditions — Pseudomonas Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Isolation of anti-Pseudomonas antibodies from type B lymphocytes — Blood sampling. Isolation of mononuclear cells from human peripheral blood by density gradient centrifugation. Identification of functional anti-Pseudomonas antibodies by ELISA and cellular infection assays.

SUMMARY:
Pseudomonas aeruginosa is a pathogenic bacteria for human, especially in hospital settings. It can sometimes be multi-resistant to many or even to all antibiotics usually used for its treatment.

The aim of the study is to isolate and produce therapeutic antibodies against the bacteria Pseudomonas aeruginosa in order to provide an alternative treatment to antibiotics in case of infection with an antibiotic-resistant strain of Pseudomonas aeruginosa.

ELIGIBILITY:
Inclusion Criteria:

* Patient selected in the retrospective part of the study (patient with serum containing functional anti-Pseudomonas aeruginosa antibodies)
* Patient with weight ≥ 32kg.
* With a follow-up visit at Grenoble University Hospital with a blood sampling for its care
* Having given its written no objection to participate in the prospective phase of this project

Exclusion Criteria:

* Legally protected patient (minor, pregnant or nursing woman, ward or ward curated, hospitalized under duress or deprived of liberty)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient previously infected or colonized by Pseudomonas aeruginosa with serum containing functional anti-Pseudomonas aeruginosa antibodies
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Isolation of recombinant human monoclonal antibodies against Pseudomonas aeruginosa | 1 day
  Detection of binding of recombinant antibodies to Pseudomonas aeruginosa target proteins by ELISA assay.

SECONDARY OUTCOMES:
Isolation of functional antibodies against Pseudomonas aeruginosa | 1 day
  Percentage of inhibition of Pseudomonas aeruginosa infection by antibodies using an in vitro model of cell infection and virulence. Percentage of lysis of Pseudomonas aeruginosa in the presence of recombinant IgG, complement and macrophages in an opsonophagocytosis assay

CONTACTS AND LOCATIONS:
Overall Officials: Yvan CASPAR, Dr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DiGiandomenico A, Sellman BR. Antibacterial monoclonal antibodies: the next generation? Curr Opin Microbiol. 2015 Oct;27:78-85. doi: 10.1016/j.mib.2015.07.014. Epub 2015 Aug 25. PMID 26302478
- [Background] Czaplewski L, Bax R, Clokie M, Dawson M, Fairhead H, Fischetti VA, Foster S, Gilmore BF, Hancock RE, Harper D, Henderson IR, Hilpert K, Jones BV, Kadioglu A, Knowles D, Olafsdottir S, Payne D, Projan S, Shaunak S, Silverman J, Thomas CM, Trust TJ, Warn P, Rex JH. Alternatives to antibiotics-a pipeline portfolio review. Lancet Infect Dis. 2016 Feb;16(2):239-51. doi: 10.1016/S1473-3099(15)00466-1. Epub 2016 Jan 13. PMID 26795692
- [Background] Rappuoli R, Bottomley MJ, D'Oro U, Finco O, De Gregorio E. Reverse vaccinology 2.0: Human immunology instructs vaccine antigen design. J Exp Med. 2016 Apr 4;213(4):469-81. doi: 10.1084/jem.20151960. Epub 2016 Mar 28. PMID 27022144
- [Background] Walker LM, Huber M, Doores KJ, Falkowska E, Pejchal R, Julien JP, Wang SK, Ramos A, Chan-Hui PY, Moyle M, Mitcham JL, Hammond PW, Olsen OA, Phung P, Fling S, Wong CH, Phogat S, Wrin T, Simek MD; Protocol G Principal Investigators; Koff WC, Wilson IA, Burton DR, Poignard P. Broad neutralization coverage of HIV by multiple highly potent antibodies. Nature. 2011 Sep 22;477(7365):466-70. doi: 10.1038/nature10373. PMID 21849977
- [Background] Holzlohner P, Hanack K. Generation of Murine Monoclonal Antibodies by Hybridoma Technology. J Vis Exp. 2017 Jan 2;(119):54832. doi: 10.3791/54832. PMID 28117810